CLINICAL TRIAL: NCT05019235
Title: Study of the Association Between Tumor Microenvironment Macrophages and Treatment Response in Squamous Cell Carcinoma of the Anal Canal
Acronym: MACARAN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: MACARAN
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Squamous cell carcinoma of the anal canal is a relatively rare cancer (less than 3% of digestive cancers) but its incidence has been increasing in recent decades, probably because of its association with HPV (human papillomavirus) infection. Its extension is mainly locoregional pelvic by lymphatic route, rarely metastatic. The standard treatment nowadays is radiotherapy combined with chemotherapy for locally advanced tumors (T2 or more corresponding to a size of 2 cm or more, or N+): mitomycin C and 5-FU (or capecitabine). While the 5-year disease control rates are excellent in localized forms, around 80%, for locally advanced tumors, the prognosis is poorer, with only 70% progression-free survival at 3 years in patients treated with radiochemotherapy. In these patients, it seems particularly interesting to understand the mechanisms of tumor resistance to treatments, in order to increase their efficacy and to propose new therapeutic targets.

The microenvironment of solid tumors, which has been extensively studied in the last two decades, is now recognized as a major factor in tumor development and invasion. Immune cells, and more particularly macrophages, represent an essential component of the tumor microenvironment, and constitute a link between innate and adaptive responses. The presence of tumor-associated macrophages (TAMs), and in particular M2 macrophages, with an anti-inflammatory and anti-tumor action (as opposed to M1 macrophages which are on the contrary tumoricidal and pro-inflammatory), has been studied in many cancers, such as head and neck squamous cell carcinoma, hepatocellular carcinoma, cervical squamous cell carcinoma, and non-small cell lung cancer. To investigator's knowledge, it has not been studied in squamous cell carcinoma of the anal canal.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient with locally advanced squamous cell carcinoma of the anal canal for which he/she has received radiotherapy/chemotherapy: tumor > 2cm and/or locoregional lymph node involvement
* Patient whose main treatment (radiotherapy and chemotherapy) was performed at the Paris Saint-Joseph Hospital
* French-speaking patient

Exclusion Criteria:

* Patient with missing or unanalyzable material
* Patient with missing data
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with locally advanced squamous cell carcinoma of the anal canal for which he/she has received radiotherapy/chemotherapy: tumor > 2cm and/or locoregional lymph node involvement, whose main treatment (radiotherapy and chemotherapy) was performed at the Paris Saint-Joseph Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of tumor-associated macrophages on treatment efficacy in locally advanced | Year 1
  This outcome corresponds to tumor recurrence (local or distant) at 1 year.

SECONDARY OUTCOMES:
Phenotype of tumor-associated macrophages | Year 1
  This outcome corresponds to distribution of tumor-associated macrophages according to their phenotype, M1 or M2, and their location (intra-tumor, peri-tumor stroma).

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Raymond, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Moureau-Zabotto L, Vendrely V, Abramowitz L, Borg C, Francois E, Goere D, Huguet F, Peiffert D, Siproudhis L, Ducreux M, Bouche O. Anal cancer: French Intergroup Clinical Practice Guidelines for diagnosis, treatment and follow-up (SNFGE, FFCD, GERCOR, UNICANCER, SFCD, SFED, SFRO, SNFCP). Dig Liver Dis. 2017 Aug;49(8):831-840. doi: 10.1016/j.dld.2017.05.011. Epub 2017 May 23. PMID 28610905
- [Background] Abramowitz L, Jacquard AC, Jaroud F, Haesebaert J, Siproudhis L, Pradat P, Aynaud O, Leocmach Y, Soubeyrand B, Dachez R, Riethmuller D, Mougin C, Pretet JL, Denis F. Human papillomavirus genotype distribution in anal cancer in France: the EDiTH V study. Int J Cancer. 2011 Jul 15;129(2):433-9. doi: 10.1002/ijc.25671. Epub 2010 Nov 9. PMID 20839262
- [Background] James RD, Glynne-Jones R, Meadows HM, Cunningham D, Myint AS, Saunders MP, Maughan T, McDonald A, Essapen S, Leslie M, Falk S, Wilson C, Gollins S, Begum R, Ledermann J, Kadalayil L, Sebag-Montefiore D. Mitomycin or cisplatin chemoradiation with or without maintenance chemotherapy for treatment of squamous-cell carcinoma of the anus (ACT II): a randomised, phase 3, open-label, 2 x 2 factorial trial. Lancet Oncol. 2013 May;14(6):516-24. doi: 10.1016/S1470-2045(13)70086-X. Epub 2013 Apr 9. PMID 23578724
- [Background] Evrard D, Szturz P, Tijeras-Raballand A, Astorgues-Xerri L, Abitbol C, Paradis V, Raymond E, Albert S, Barry B, Faivre S. Macrophages in the microenvironment of head and neck cancer: potential targets for cancer therapy. Oral Oncol. 2019 Jan;88:29-38. doi: 10.1016/j.oraloncology.2018.10.040. Epub 2018 Nov 20. PMID 30616794
- [Background] Cao L, Che X, Qiu X, Li Z, Yang B, Wang S, Hou K, Fan Y, Qu X, Liu Y. M2 macrophage infiltration into tumor islets leads to poor prognosis in non-small-cell lung cancer. Cancer Manag Res. 2019 Jul 4;11:6125-6138. doi: 10.2147/CMAR.S199832. eCollection 2019. PMID 31308749